CLINICAL TRIAL: NCT03665935
Title: Role of Diffusion Tensor Imaging in Evaluation of Myelopathy
Brief Title: Diffusion Tensor Imaging of Myelopathy
Acronym: DTI
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, MGMaghrabi, principle investigator, Assiut University
Other Study IDs: DTI in myelopathy
Record Dates: First submitted 2018-09-06; First posted 2018-09-11 (Actual); Last update posted 2018-09-11 (Actual); Status verified 2018-09

CONDITIONS: Myelopathy
MeSH Terms: conditions — Spinal Cord Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Myelopathy describes any neurologic deficit related to the spinal cord. Myelopathy is caused by various pathological states of the human spinal cord, including tumors, inflammatory lesions, spinal cord compression and degenerative myelopathy. Clinically, the diagnosis of myelopathy depends on localization of the neurologic finding to the spinal cord, rather than the brain or peripheral nervous system and then to a particular segment of the spinal cord.

Magnetic resonance imaging (MRI) plays an essential role in the diagnosis and follow-up of the lesions of the spinal cord using conventional MRI T1- and T2-weighted sequences. Sometimes a studied spinal cord may appear normal on conventional MRI even though patients have symptoms of myelopathy causing a discrepancy between MRI findings and clinical findings.

Diffusion tensor imaging (DTI) is an advanced non-invasive MR imaging technique which assesses the microstructural integrity of nerve fiber tracts.

DETAILED DESCRIPTION:
A number of 70 patient with myelopathy included within the study.

DTI is used primarily for assessing white matter of the brain and spinal cord. DTI can depict alterations to the white matter tract and quantify these changes. Disturbances of diffusion (restriction or increase) may be assessed quantitatively by measurements of apparent diffusion coefficient (ADC). The apparent diffusion coefficient (ADC), is used to measure diffusive strength. Diffusion anisotropy can be assessed quantitatively by using the fractional anisotropy (FA) parameter, which may be also visualized on fractional anisotropy maps. FA is considered as a marker of white matter integrity.

Image acquisition will be conducted on a 1.5-Tesla MR scanner.

The imaging will be done throughout the following sequences:

1. Conventional MRI sequences: sagittal T1W, sagittal and axial T2W sequences.
2. DTI sequence: Single-shot spin-echo echo-planar imaging (EPI) and parallel imaging techniques to achieve motion-free and higher signal-to-noise ratio (SNR) DTI.

Post processing:

The diffusion-tensor imaging data is transferred to an offline workstation utilizing software used for reconstruction of the Diffusion Tensor imaging (DTI) with regions of interest were defined and measured on the ADC and fractional anisotropy (FA) maps. diffusion tensor tractogram will be constructed on the acquired data source.

ELIGIBILITY:
Inclusion Criteria:

* Clinical symptoms of myelopathy

Exclusion Criteria:

* Previous spine surgery
* Spine radiation therapy
* Cerebral palsy
* Contraindication to MR imaging.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: A 70 patient with myelopathy will be included in the study. the study will be performed at radiology department in Assiut University Hospital. Using Magnetic Resonance imaging device 1.5 tesla scanners. First imaging the spine by acquiring the conventional sequences and second the diffusion tensor sequence.
Sampling Method: Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2018-09 (Estimated); Primary Completion 2019-09 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
To determine the usefulness of diffusion tensor imaging (DTI) and fiber tracking in evaluation of myelopathy. | one year
  assessing white matter tract affection in various disease and damage involving the spinal cord using the DTI indices, quantitatively using ADC and FA measurement and qualitatively using tractogram to assess spinal cord lesions and compare the results to conventional MRI sequences

CONTACTS AND LOCATIONS:
Overall Officials: Mona Gouda, ass lecturer, Principal Investigator — Assiut University

REFERENCES:
- [Background] Kamble RB, Venkataramana NK, Naik AL, Rao SV. Diffusion tensor imaging in spinal cord injury. Indian J Radiol Imaging. 2011 Jul;21(3):221-4. doi: 10.4103/0971-3026.85372. PMID 22013299